CLINICAL TRIAL: NCT02558140
Title: An Open-Label, Multicenter, Dose-Escalation Phase I Study of RO6874813, Administered Intravenously in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Dose Escalation Study of RO6874813 in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP29773; RG7386 (Other: Roche); 2015-001889-26 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-23 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation (Experimental): All participants will be given RO6874813 as a single low dose of 0.5 milligrams per kilogram (mg/kg) via intravenous (IV) infusion in a 7-day pharmacokinetic (PK) run-in period (Cycle 0). This is followed by dose escalation (Cycle 1) for which participants will receive escalating doses of RO6874813 (starting dose = 1 mg/kg) via IV infusion every week (qw) or every 2 weeks (Q2W) for 28 to 42 days to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D).
  Interventions: Biological: RO6874813
- Part 2: Tumor Biopsy and Imaging (Experimental): The first 15 participants with fibroblast activation protein-alpha positive (FAP+) tumors will be treated at the RP2D and dosing schedule as determined in Part 1, and will undergo paired tumor biopsies for biomarker assessments. Up to 5 participants with FAP+ tumors will undergo baseline and on-treatment tumor biopsies for biomarker assessments at a dose below the RP2D. The dose for these participants can be escalated to RP2D after 4 weeks of treatment and upon completion of biomarker assessment.
  Interventions: Biological: RO6874813
- Part 3: Preliminary Efficacy Assessment (Experimental): Participants with locally advanced or metastatic non-resectable FAP+ sarcoma will be treated with RO6874813 at the RP2D and as per schedule determined upon completion of Part 1. Participants continuing treatment with RO6874813 beyond 36 weeks will enter the extension phase of Part 3 and will be monitored for disease status and clinical safety per routine standard of care.
  Interventions: Biological: RO6874813

INTERVENTIONS:
Biological: RO6874813 — RO6874813 will be administered at a single low dose of 0.5 mg/kg via IV infusion in a 7- day PK run-in period (Cycle 0). Dose level for RO6874813 will be escalated to determine MTD and RP2D for RO6874813.
  Arms: Part 1: Dose Escalation
Biological: RO6874813 — RO6874813 at RP2D will be administered by IV infusion as per dosing schedule determined in Part 1.
  Arms: Part 2: Tumor Biopsy and Imaging; Part 3: Preliminary Efficacy Assessment

SUMMARY:
This first-in-human study consists of three parts. The primary purpose of Part 1 is to characterize the safety and tolerability of RO6874813 in participants with locally advanced and/or metastatic solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists. In addition, the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) will be determined. In Part 2 the safety and tolerability of RO6874813 will continue to be characterized in participants with locally advanced and/or metastatic solid tumors known to be fibroblast activation protein-alpha positive (FAP+). In addition, treatment-induced efficacy of RO6874813 will be assessed by functional imaging and paired tumor biopsies. The primary purpose of Part 3 is to demonstrate anti-tumor activity of RO6874813 in participants with recurrent or metastatic FAP+ sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Participants with histologically/cytologically confirmed locally advanced or metastatic, non-resectable solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists
* Part 2: Participants with histologically/ cytologically confirmed locally advanced or metastatic, non-resectable solid tumors known to be FAP+ whose disease has progressed despite standard therapy or for whom no standard therapy exists
* Part 3: Participants with histologically confirmed recurrent or metastatic, non-resectable confirmed FAP+ sarcoma with two or fewer prior regimens for advanced disease
* All participants must have tumor tissue that can be imaged for pharmacodynamic assessments and from which a pre- and on-treatment biopsy can be safely obtained
* An archival tumor sample must be available for retrospective FAP expression analysis
* Measurable disease as determined by RECIST v1.1
* World Health Organization (WHO)/ Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
* Recovery from all reversible AEs of previous anti-cancer therapies to baseline or Common Terminology Criteria for Adverse Events (CTCAE) Grade 1, except for alopecia (any grade) and Grade <=2 sensory peripheral neuropathy
* Negative pregnancy test

Exclusion Criteria:

* Primary central nervous (CNS) tumors or CNS tumor involvement
* Major surgery or any other prior anti-cancer treatment within 4 weeks prior to study Day 1.
* Received wide-field radiotherapy <= 4 weeks or limited-field radiotherapy <=2 weeks prior to starting study drug
* Known hypersensitivity to any of the components of RO6874813 or to the contrast agents used in the study
* Another invasive malignancy in the last 2 years except for those with a minimal risk of metastasis or death
* Any other conditions or diseases that would contraindicate participation in the clinical study because of safety concerns or compliance with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10-11 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants With Dose-Limiting Toxicity (DLT) | 28 days
Part 1: Maximum Tolerated Dose (MTD) of RO6874813 | 28 days
Part 1: Recommended Phase 2 Dose (RP2D) of RO6874813 | 28 days
Parts 1 and 2: Percentage of Participants With Adverse Events (AEs) | Baseline up to approximately 24 months
Parts 1 and 2: Percentage of Participants With Anti-Drug Antibodies (ADAs) | Predose (Hour [Hr] 0) on Day 1 up to approximately 12 months; please see outcome measure description for detailed time frame
  Q2W (1 cycle=14 days): Predose (Hr 0) on Day 1 of Run-in period (Part 1 only), Cycles 1, 3, 5, then every 2 cycles (up to approximately 12 months); QW (1 cycle=7 days): Predose on Day 1 of Run-in period (Part 1 only), Cycles 1, 2, 5, then every 2 cycles (up to approximately 12 months)
Part 3: Percentage of Participants With Objective Response as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Baseline until disease progression (up to approximately 12 months)
Part 3: Percentage of Participants With Disease Control as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 3: Duration of Response (DoR) as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 3: Median Progression-Free Survival (PFS) as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 3: Percentage of Participants Who are Progression-Free at Months 3 as Determined by the Investigator Using RECIST v1.1 | Month 3
Part 3: Percentage of Participants Who are Progression-Free at Month 6 as Determined by the Investigator Using RECIST v1.1 | Month 6
Part 3: Median Overall Survival (OS) | Baseline until death (up to approximately 24 months)
Part 3: Percentage of Participants Who are Alive at Month 12 | Month 12

SECONDARY OUTCOMES:
Parts 1, 2, and 3: Maximum Observed Serum Concentration (Cmax) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), End of Infusion (EoI) (infusion length less than or equal to [<=] 1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Minimum Observed Serum Concentration (Cmin) of RO6874813 | QW or Q2W: Predose (Hr 0) on Day 1 in Cycles 0, 1, 2, 3, 4, 5, 6, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Time to Reach Cmax (Tmax) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), EoI (infusion length <=1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Half-Life (t1/2) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), EoI (infusion length <=1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Area Under the Concentration-Time Curve (AUC) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), EoI (infusion length <=1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Clearance (CL) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), EoI (infusion length <=1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: AUC During One Dose Interval (AUCtau) of RO6874813 | Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycle 1 and QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycle 1
Parts 1, 2, and 3: Volume at Steady State (Vss) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), EoI (infusion length <=1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Accumulation Ratio (RA) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Run-in Period (Part 1 only): Predose (Hr 0), EoI (infusion length <=1.5 hrs), 24, 48, 72 (only for QW), and 96 hrs after EoI. Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose and EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months). QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycles 1 and 4; Predose, EoI, and 2 hrs after EoI in Cycles 2 and 6; Predose, EoI in Cycles 3, 5, 7, and every 2 cycles thereafter (up to approximately 12 months)
Parts 1, 2, and 3: Observed Steady-State Concentration at the End of a Dosing Interval (Ctrough) of RO6874813 | Predose (Hr 0) up to approximately 12 months; please see outcome measure description for detailed time frame
  Q2W (1 cycle=14 days): Predose, EoI, 2, 6, 24, 72, 96, 168, and 240 hrs after EoI in Cycle 1. QW (1 cycle=7 days): Predose, EoI, 2, 6, 24, 48, 72, and 96 hrs after EoI in Cycle 1
Parts 1, 2, and 3: Change from Baseline in Body Weight Corrected Maximum Standardized Uptake Volume (SUVmax) as Measured by 2-[18F]Fluoro-2-Deoxyglucose Positron Emission Tomography ([18F]-FDG PET) | Baseline and 12 months
Part 1 and 2: Percentage of Participants With Objective Response as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 1 and 2: Percentage of Participants With Disease Control as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 1 and 2: DOR as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 1 and 2: Median PFS as Determined by the Investigator Using RECIST v1.1 | Baseline up to approximately 12 months
Part 1 and 2: Percentage of Participants Who are Progression-Free at Month 6 as Determined by the Investigator Using RECIST v1.1 | Month 6
Part 3: Percentage of Participants With AEs | Baseline up to approximately 24 months
Part 3: Percentage of Participants With ADAs | Predose (Hr 0) on Day 1 up to approximately 12 months; please see outcome measure description for detailed time frame
  Q2W (1 cycle=14 days): Predose (Hr 0) on Day 1 of Run-in period (Part 1 only), Cycles 1, 3, 5, then every 2 cycles (up to approximately 12 months); QW (1 cycle=7 days): Predose on Day 1 of Run-in period (Part 1 only), Cycles 1, 2, 5, then every 2 cycles (up to approximately 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- SCRI, Nashville, Tennessee, United States
- Centre Leon Berard; Departement Oncologie Medicale, Lyon, France
- Spain (2):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid